CLINICAL TRIAL: NCT02169115
Title: Double-blind, Placebo-controlled 12-week, Parallel-group Study With a 6 Weeks Follow up Period to Demonstrate Efficacy and Safety of Subcutaneous Omalizumab in Patients With Urticaria Factitia Refractory to Standard Treatment
Brief Title: Urticaria Facticia Treatment With Omalizumab (UFO)
Acronym: UFO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Martin Metz, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025EDE17T; 2011-005615-87 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Symptomatic Dermographism
MeSH Terms: conditions — Familial dermographism | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omalizumab 150mg (Experimental)
  Interventions: Drug: Omalizumab
- Omalizumab 300mg (Experimental)
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — 150mg, s.c., every 4 weeks
  Other Names: Xolair
  Arms: Omalizumab 150mg
Drug: Omalizumab — 300mg, s.c., every 4 weeks
  Other Names: Xolair
  Arms: Omalizumab 300mg
Drug: Placebo — Placebo, s.c., every 4 weeks
  Arms: Placebo

SUMMARY:
Urticaria is a very frequent skin condition characterized by transient wheal and flare type skin reactions associated with severe pruritus. In Europe alone, more than 5 million patients are thought to suffer from persisting urticaria symptoms, which either occur spontaneously, i.e. in chronic spontaneous urticaria (CSU), or as a result of environmental physical stimuli such as friction, pressure, UV irradiation or cold (physical urticaria). Urticaria factitia (also known as dermographic urticaria and symptomatic dermographism) is characterized by whealing and itching following a minor stroking pressure, rubbing or scratching of the skin. The majority of patients with urticaria factitia benefits from treatment with nonsedating antihistamines. Some patients, however, do not achieve adequate symptom control even with updosing of antihistamines and may suffer from substantial quality of life impairment . Since even very minor stroking of the skin can lead to the development of wheals and severe itching, these patients are for example limited in their choice of clothing and are impaired in their social interaction and partnership.

In all patients with a history of wheals after stroking of the skin, a provocation test should be performed. This can be done by stroking of the skin lightly with a smooth blunt object (e.g. the tip of a closed ball point pen or a wooden spatula) or a purpose-built instrument, known as a dermographometer. For the diagnosis of symptomatic dermographism, the smooth blunt object should be held perpendicular to the skin and should be used to apply a light stroking pressure to the skin of the upper back or volar forearm. The reaction is considered positive in patients who show a weal response and report pruritus at the site of provocation.

Patients with a positive test reaction should be evaluated for individual pressure thresholds. For this purpose a provocation device (FricTest) has been developed that allows for reproducible and standardized threshold testing. Threshold testing enables physicians to assess disease severity and treatment response more precisely.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-75 years)
* Informed consent signed and dated
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Diagnosis of UF lasting for at least 6 months
* Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to have SC injections administered by a qualified person
* In females of childbearing potential: Negative pregnancy test; females willing to use highly effective contraception (Pearl-Index < 1). A woman will be considered not of childbearing potential if she is post-menopausal for greater than two years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion Criteria:

* Patients with acute urticaria
* Concurrent/ongoing treatment with immunosuppressives (e.g. systemic steroids, cyclosporine, methotrexate, dapsone or others) within 4 weeks or 5 half lives prior to day 0, whichever is longer
* Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial
* Significant concomitant illness that would adversely affect the subject's participation or evaluation in this study
* History of malignancies within five years prior to screening other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cancer
* Presence of clinically significant laboratory abnormalities
* Lactating females or pregnant females
* Subjects for whom there is concern about compliance with the protocol procedures
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk
* History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) within the last 5 years that could limit the subject's ability to comply with study procedures
* Subjects who are detained officially or legally to an official institute
* Previous use of omalizumab within the last 6 months
* Intake of antihistamines or leukotriene antagonists within 4 days prior to visit 1
* Intake of oral corticosteroids within 14 days prior to visit 1
* Use of depot corticosteroids or chronic systemic corticosteroids within 21 days before beginning of the study
* Known hypersensitivity to any ingredients, including excipients (sucrose, histidine, polysorbate 20) of the study medication or drugs related to omalizumab (e.g.: monoclonal antibodies, polyclonal gammaglobulin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Metz, MD, Principal Investigator — Charité University
Locations (2):
- Germany (2):
  - University Dermatology Freiburg, Freiburg im Breisgau
  - Dermatology University Mainz, Mainz

REFERENCES:
- [Derived] Maurer M, Schutz A, Weller K, Schoepke N, Peveling-Oberhag A, Staubach P, Muller S, Jakob T, Metz M. Omalizumab is effective in symptomatic dermographism-results of a randomized placebo-controlled trial. J Allergy Clin Immunol. 2017 Sep;140(3):870-873.e5. doi: 10.1016/j.jaci.2017.01.042. Epub 2017 Apr 4. No abstract available. PMID 28389391

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Started | 19 | 21 | 21
Completed | 19 | 21 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 21 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 21 | 61
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 12 | 34
  Male | 6 | 12 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Germany | 19 | 21 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Provocation Thresholds From Baseline to Day 70 in Urticaria Factitia Patients After Treatment With Omalizumab Compared to Placebo
Description: Patients receive provocation test by FricTest (standardized stroking of the skin). FricTest ratings are from 0 (no wheal development to the longest pin) to 4 (wheal development to all four pins). The development of wheals within 30 minutes after provocation is monitored.
Time Frame: 70 days
Measure: Mean (Standard Deviation); unit: wheal development up to four pins
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
wheal development up to four pins | -1.8 (1.7) | -2.0 (1.8) | -0.6 (1.4)
Statistical Analysis 1: Comparison: Omalizumab 150mg; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Final Values) = -1.8, Standard Deviation 1.7
Statistical Analysis 2: Comparison: Omalizumab 300mg; Test type: Superiority or Other; p = 0.005, ANOVA; Mean Difference (Final Values) = 2.0, Standard Deviation 1.8
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, Standard Deviation 1.4

2. Secondary Outcome: To Assess the Effects of Omalizumab in Urticaria Factitia Patients on Quality of Life
Description: Change in quality of life scores assessed by Dermatology Life Quality Index (DLQI) and UF specific life quality questions from baseline to day 70 after treatment with omalizumab compared to placebo. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percantage of the maximum possible score of 30.
Time Frame: 70 days
Measure: Mean (Standard Error); unit: Dermatology quality of life score
Groups:
- Placebo: Placebo: s.c., every 4 weeks
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
Dermatology quality of life score | -6.611 (1.234) | -5.579 (1.478) | -2.316 (0.949)

3. Secondary Outcome: To Assess the Effects of Omalizumab in UF Patients on Number of Symptom Free Days
Description: Change in number of symptom free days as assessed by a patient diary from baseline to day 70 after treatment with omalizumab compared to placebo
Time Frame: 70 days
Population: Data were not collected.
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: To Assess the Effects of Omalizumab in UF Patients on Physician Global Assessment of Disease Severity
Description: Change in physician global assessment of disease severity assessed by visual analogue scale by a physician from baseline to day 70 after treatment with omalizumab compared to placebo. VAS are measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients. The scale ranges from a minimum of 0 and a maximum of 10. The higher the score, the worse the outcome.
Time Frame: 70 days
Measure: Mean (Standard Error); unit: units on a sclae
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 18 | 19 | 20
units on a sclae | 21.8 (3.63) | 28.33 (6.23) | 40.32 (6.162)

5. Secondary Outcome: To Assess the Effects of Omalizumab in UF Patients on Patient Global Assessment of Disease Severity
Description: Change in patient global assessment of disease severity assessed by visual analogue scale by the patient from baseline to day 70 after treatment with omalizumab compared to placebo. VAS are measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients. The scale ranges from a minimum of 0 and a maximum of 10. The higher the score, the worse the outcome.
Time Frame: 70 days
Population: Data were not collected.
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: To Assess Long-term Effects of Omalizumab in UF Patients
Description: To assess long-term effects of omalizumab in UF patients, change in friction thresholds from day 70 (week 10) to day 112 (week 16) will be assessed
Time Frame: 112 days
Measure: Mean (Standard Deviation); unit: Fric Test grades
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 18 | 19 | 18
Fric Test grades | -1.0556 (1.39209) | -0.8421 (1.77210) | -0.8333 (1.50489)

7. Secondary Outcome: Number of Participants With Serious Adverse Events and Adverse Events
Description: Safety of patients treated with omalizumab: This includes physical examination, routine safety laboratory assessments, vital signs and adverse event reporting
Time Frame: 112 days
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Number analyzed (Participants) | 19 | 21 | 21
Participants
  Patients with serious adverse events | 1 | 1 | 1
  Patients with adverse events | 17 | 17 | 19

ADVERSE EVENTS:
Arm/Group | Omalizumab 150mg | Omalizumab 300mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 18/19 | 15/21 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 150mg (N=19) | Omalizumab 300mg (N=21) | Placebo (N=21)
inguinal hernia (Surgical and medical procedures) | 1 | 0 | 0
Unspecified renal colic (Renal and urinary disorders) | 0 | 0 | 1
Acute cystitis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 150mg (N=19) | Omalizumab 300mg (N=21) | Placebo (N=21)
Headache (General disorders) | 6 | 9 | 10
Upper respiratory tract (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No